CLINICAL TRIAL: NCT04127227
Title: Sintilimab With P-GemOx (Pegaspargase, Gemcitabine and Oxaliplatin) Regimen for Newly Diagnosed Advanced Extranodal Natural Killer/T-cell Lymphoma, Nasal Type (ENKTL): a Single Arm, Open, Multicenter, Phase II Study
Brief Title: Sintilimab With P-GemOx Regimen for Newly Diagnosed Advanced Extranodal Natural Killer/T-cell Lymphoma, Nasal Type
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-148
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: NK/T Cell Lymphoma Nos
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab With P-GemOx (Experimental): Sintilimab, 200mg, d1, intravenous drip; pegaspargase, 2000U/m2, d1, intravenous drip; gemcitabine, 1000mg/m2, d1,d8, intravenous drip; oxaliplatin, 130mg/m2, d1, intravenous drip; All patients received up to 6 treatment cycles of 21 days. Patients with CR or PR will receive Sintilimab maintenance therapy.
  Interventions: Drug: sintilimab,pegaspargase,gemcitabine,oxaliplatin

INTERVENTIONS:
Drug: sintilimab,pegaspargase,gemcitabine,oxaliplatin — All patients enrolled in the study will accept sintilimab with P-GemOx (pegaspargase, gemcitabine and oxaliplatin) regimens their first-line therapy.
  Patients with CR or PR will receive sintilimab maintenance therapy

SUMMARY:
The purpose of this multi-center,single arm,phase Ⅱ clinical trail is to determine the safety and efficacy of Sintilimab with P-GemOx (pegaspargase, gemcitabine and oxaliplatin) regimen for newly diagnosed advanced extranodal natural killer/T-cell lymphoma, nasal type (ENKTL)

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved extranodal natural killer/T-cell lymphoma, nasal type;
* newly diagnosed stage III/IV patients;
* at least one evaluable lesion；
* ECOG PS 0-2;
* 18-75 years; without other malignancy;
* proper functioning of the major organs.

Exclusion Criteria:

* hemophagocytic syndrome or aggressive NK cell leukemia;
* involvement of central nervous system;
* previously received treatment of chemotherapy, radiotherapy, immunotherapy or biotherapy for lymphoma；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2023-10-09 (Estimated); Study Completion 2023-10-09 (Estimated)

PRIMARY OUTCOMES:
complete remission (CR) rate | 2years
overall response rate (ORR) | 2years

SECONDARY OUTCOMES:
overall survival (OS) | 2years
progression survival (PFS) | 2years
disease-free survival (DFS) | 2years
bio-marker analysis | 2years
  Correlation between programmed death-ligand 1 expression and efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Tian XP, Cai J, Xia Y, Zhang YC, Wang L, Liu PP, Huang HQ, Li YJ, Zhou H, Li ZM, Yang J, Wei LQ, Zou QH, Huang Y, Li J, Ling L, Zhong WL, Cai QQ. First-line sintilimab with pegaspargase, gemcitabine, and oxaliplatin in advanced extranodal natural killer/T cell lymphoma (SPIRIT): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2024 May;11(5):e336-e344. doi: 10.1016/S2352-3026(24)00066-8. Epub 2024 Mar 27. PMID 38554717